CLINICAL TRIAL: NCT04093908
Title: Machine Learning Prediction of Motor Response After STN DBS in Parkinson Patients, a Retrospective Multicenter Validation Study
Brief Title: Prediction of STN DBS Motor Response in PD
Acronym: DBS-PREDICT
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0739-A9
Record Dates: First submitted 2019-09-17; First posted 2019-09-18 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
Keywords: deep brain stimulation; motor outcome; prediction model; machine learning; Subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multi-center validation cohort: We collect retrospective data from several international centers containing preoperative variables (demographical and clinical) and postoperative outcome (UPDRS II, III, IV) one year postoperatively, and merge these data to one validation cohort.
  Interventions: Other: Prediction of motor outcome after STN DBS based on preoperative variables

INTERVENTIONS:
Other: Prediction of motor outcome after STN DBS based on preoperative variables — Generating individual probabilities for motor response based on preoperative variables

SUMMARY:
Despite careful patient selection for subthalamic nucleus deep brain stimulation (STN DBS), some Parkinson's disease (PD) patients show limited improvement of motor disability. Non-conclusive results and the lack of a practical implantable prediction algorithm from previous prediction studies maintain the need for a simple tool for neurologists that provides a reliable prediction on postoperative motor improvement for individual patients.

In this study, a prior developed prediction model for motor response after STN DBS in PD patients is validated. The model generates individual probabilities for becoming a weak responder one year after surgery. The model will be validated in a validation cohort collected from several international centers.

The predictive model is made public accessible before data collection on: https://github.com/jgvhabets/DBSPREDICT

DETAILED DESCRIPTION:
Predicting motor outcome after STN DBS in Parkinson Disease can be challenging for the clinician. Current prediction studies report non-conclusive results on the most important predictors and are limited by used computational methods. Traditional statistical analyses which focus on correlations are biased by predictor- and confounder-selection by the investigators. Modern computational methods like machine learning prediction models are less limited by sample size and can consider a wider range of predictors which leads to less selection-bias.

Retrospective patient data is collected from multiple international centers. This retrospective, multicenter cohort is used to validate the model which is developed based on a single-center retrospective cohort.

The goal is to develop a prediction tool that provides the clinician with a probability for weak response during the preoperative phase. This could support the clinician in including or informing the patient during preoperative counseling.

The predictive model is made public accessible before data collection on: https://github.com/jgvhabets/DBSPREDICT.

ELIGIBILITY:
Inclusion Criteria:

* underwent STN DBS for Parkinson's disease
* completed one year follow up after surgery

Exclusion Criteria:

- missing data in postoperative UPDRS II, III, IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One cohort consisting of PD patients who underwent STN DBS in several international centers.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
area under the curve of the receiver operator curve | one-year postoperative
  Motor outcome is categorised in a binary outcome variable. The model will predict to which outcome group the patient will belong one-year postoperatively. The primary outcome measure is the performance of the predicted outcome categories with the actual outcome categories.
  Performance of prediction models is expressed as area under the curve of the receiver operator curve, predictive accuracy, true positive prediction rate, and false positive prediction rate.
predictive accuracy | one-year postoperative
  See description primary outcome 1.
true positive prediction rate | one-year postoperative
  See description primary outcome 1.
false positive prediction rate | one-year postoperative
  See description primary outcome 1.

CONTACTS AND LOCATIONS:
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared after completing analysing
Supporting Information: Study Protocol, Analytic Code
Time Frame: After data collection and analysis.
Access Criteria: Data can be made available on request.